CLINICAL TRIAL: NCT06820671
Title: Voice Analysis in Asthmatic Patients and Healthy Individuals: Comparative Evaluation of Asthma Control Levels and Voice Characteristics With Machine Learning Models
Brief Title: Voice Analysis in Asthmatic Patients With Machine Learning Models
Status: Completed | Type: Observational
Sponsor: MED-CASE (Other)
Collaborators: Saglik Bilimleri Universitesi (Other); Yedikule Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Med-ML001
Record Dates: First submitted 2025-01-15; First posted 2025-02-11 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Asthma
Keywords: voice biomarker; machine learning
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Asthmatic Group: Diagnosed asthma patients Adults aged between 18 and 65 years of age who have been diagnosed with asthma and followed-up for at least 3 months
  Interventions: Other: Recording voice samples
- Healthy Group: Healthy participants Adults aged between 18-65 years of age with good general health
  Interventions: Other: Recording voice samples

INTERVENTIONS:
Other: Recording voice samples — Voice recording with
  * reading the standard text
  * repeating the test words
  * vowel elicitation of 'a' and 'o' vowels for 5-10 seconds

SUMMARY:
Asthma can lead to various factors that impair voice production, including airway restriction, inflammation, and mucus production, resulting in changes in voice frequency and amplitude. Therefore, voice analysis may serve as an indicator of respiratory diseases.

A national, observational, case-control study is planned in Türkiye to analyze differences in voice between healthy subjects and asthmatic patients and to assess voice analysis techniques for determining an effective biomarker for asthma control using a machine learning model.

DETAILED DESCRIPTION:
Asthma is a disease characterized by chronic inflammation. Based on the frequency of symptoms and the use of reliever medications, the disease can be classified as either 'controlled' or 'uncontrolled'. Currently, GINA criteria and Asthma Control Test can be used to evaluate asthma control.

The relationship between respiratory functions and speech has been previously studied, revealing that voice changes can occur in asthmatic patients due to symptom presence. Asthma can lead to various factors that impair voice production, including airway restriction, inflammation, and mucus production, resulting in changes in voice frequency and amplitude. Therefore, voice analysis may serve as an indicator of respiratory diseases. Understanding the alterations in phonation/voice due to the underlying disease is crucial.

This study seeks to analyze differences in voice between healthy subjects and asthmatic patients and to assess voice analysis techniques for determining an effective biomarker for asthma control using a machine learning model.

This is a national, observational, cross-sectional study that will be conducted in Türkiye. The study consists of two stages: in the first stage, a machine learning (ML) model will be developed using voice data collected from both healthy individuals and patients diagnosed with asthma. In the second stage, this ML model will be tested to detect voice differences among patients at different levels of asthma control.

ELIGIBILITY:
Asthmatic Group

Inclusion Criteria:

* Patients diagnosed with asthma according to GINA criteria and Pulmonary Function Test, and followed for at least three months
* 18-65 years of age.
* Sign an informed consent document
* Able to comply with the study protocol during the study period.

Exclusion Criteria:

* None

Healthy Group

Inclusion Criteria:

* Healthy participants between 18-65 years of age
* Good general health
* No history of chronic respiratory disorders
* No history of chronic systemic disorders
* No history of upper respiratory tract infections within five days prior voice recording.

Exclusion Criteria:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who admitted at Yedikule Chest Diseases and Thoracic Surgery Training And Research Hospital who meet eligibility criteria will be enrolled for 'Asthmatic Group'.
  Healthy relatives of the patients and other healthy individuals at the hospital will be enrolled for 'Healthy Group'.
Sampling Method: Non-Probability Sample
Enrollment: 344 (Actual)
Dates: Start 2024-01-09 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Comparison of voice characteristics | One session, a maximum of 7 voice sample recording in one session for each participant, 2 minutes total.
  Comparison of voice characteristics in asthmatic patients and healthy individuals with machine learning and deep learning

SECONDARY OUTCOMES:
Classification of voice characteristics | A maximum of 7 voice sample recording in one session for each participant, 2 minutes total.
  Classification of voice characteristics according to Global Initiative for Asthma - (GINA) criteria using machine learning and deep learning

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Yedikule Chest Diseases and Thoracic Surgery Training And Reseaerch Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No